CLINICAL TRIAL: NCT01457352
Title: Efficacy and Safety of SPARC0921 in Subjects With Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLR_09_21
Record Dates: First submitted 2011-10-17; First posted 2011-10-21 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Spasticity
Keywords: spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPARC0921 (Experimental)
  Interventions: Drug: SPARC0921
- Placebo0921 (Placebo Comparator)
  Interventions: Drug: Placebo0921

INTERVENTIONS:
Drug: SPARC0921
  Arms: SPARC0921
Drug: Placebo0921
  Arms: Placebo0921

SUMMARY:
The purpose of this study is to assess whether SPARC0921 demonstrate efficacy and safety in the treatment of spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years and older
* Able and willing to comply with the protocol, including availability for a scheduled clinic visits
* Willingness and giving of written informed consent

Exclusion Criteria:

* In relapse or history of unstable course over the prior 30 days prior to the Screening Visit
* Concomitant neurologic conditions causing spasticity
* Has received an investigational drug or device within 30 days that would interfere with the study goals prior to the Screening Visit
* Unable to comply with study procedures in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (56):
  - SPARC site 6, Gilbert, Arizona
  - SPARC Site 40, Phoenix, Arizona
  - SPARC Site 36, Costa Mesa, California
  - SPARC Site 20, Newport Beach, California
  - SPARC Site 38, Basalt, Colorado
  - SPARC Site 21, Denver, Colorado
  - SPARC Site 9, Derby, Connecticut
  - SPARC Site 57, Hartford, Connecticut
  - SPARC Site 10, New London, Connecticut
  - SPARC Site 60, Washington D.C., District of Columbia
  - SPARC Site 15, Bradenton, Florida
  - SPARC Site 54, Jacksonville, Florida
  - SPARC Site 41, Maitland, Florida
  - SPARC Site 70, Miami, Florida
  - SPARC Site 8, Ormond Beach, Florida
  - SPARC Site 17, Port Charlotte, Florida
  - SPARC Site 19, Sarasota, Florida
  - SPARC Site 31, Sunrise, Florida
  - SPARC Site 39, Tampa, Florida
  - SPARC Site 65, Tampa, Florida
  - SPARC Site 51, Lenexa, Kansas
  - SPARC Site 30, Overland Park, Kansas
  - SPARC Site 50, Louisville, Kentucky
  - SPARC Site 42, Alexandria, Louisiana
  - SPARC Site 27, Baton Rouge, Louisiana
  - SPARC Site 73, New Orleans, Louisiana
  - SPARC Site 35, Foxborough, Massachusetts
  - SPARC Site 23, Springfield, Massachusetts
  - SPARC Site 32, Clinton Township, Michigan
  - SPARC Site 64, Detroit, Michigan
  - SPARC Site 25, Golden Valley, Minnesota
  - SPARC Site 5, Henderson, Nevada
  - SPARC site 34, Flemington, New Jersey
  - SPARC Site 55, Stratford, New Jersey
  - SPARC Site 22, Albuquerque, New Mexico
  - SPARC Site 49, Rochester, New York
  - SPARC Site 45, Charlotte, North Carolina
  - SPARC Site 4, Charlotte, North Carolina
  - SPARC Site 24, Greensboro, North Carolina
  - SPARC Site 2, Winston-Salem, North Carolina
  - SPARC Site 75, Winston-Salem, North Carolina
  - SPARC Site 16, Akron, Ohio
  - SPARC Site 33, Centerville, Ohio
  - SPARC Site 56, Columbus, Ohio
  - SPARC Site 12, Eugene, Oregon
  - SPARC Site 44, Springfield, Oregon
  - SPARC Site 68, Abington, Pennsylvania
  - SPARC Site 29, Old Point Station, South Carolina
  - SPARC Site 7, Austin, Texas
  - SPARC Site 71, Dallas, Texas
  - SPARC Site 43, Houston, Texas
  - SPARC Site 13, Salt Lake City, Utah
  - SPARC Site 26, Tacoma, Washington
  - SPARC Site 74, Huntington, West Virginia
  - SPARC Site 69, Milwaukee, Wisconsin
  - SPARC Site 67, Waukesha, Wisconsin
- Germany (4):
  - SPARC Site 77, Dresden
  - SPARC Site 76, Erbach im Odenwald
  - SPARC Site 79, Teupitz
  - SPARC Site 78, Westerstede
- Hungary (4):
  - SPARC Site 82, Budapest
  - SPARC site 83, Budapest
  - SPARC Site 81, Eger
  - SPARC Site 80, Esztergom
- Russia (5):
  - SPARC Site 87, Moscow
  - SPARC Site 86, Novosibirsk
  - SPARC Site 85, Saint Petersburg
  - SPARC Site 84, Sestroretsk
  - SPARC Site 88, Stavropol
- Ukraine (4):
  - SPARC Site 90, Dnipropetrovsk
  - SPARC Site 92, Lviv
  - SPARC Site 91, Poltava
  - SPARC Site 89, Zaporozh’ye

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in part 1, 2, and 3:
  Part 1: 392 subjects Part 2: 376 subjects (SPARC0921), one death occurred in Part 2 of the study. Part 3: 296 subjects (SPARC0921 or Placebo0921)
  Efficacy results are presented for Part 3 and safety results are presented for Part 2 and Part 3 of the study as per the objectives of the study.
Groups:
- SPARC0921: once, twice, thrice, or four times daily for one week
- Placebo: Placebo formulation
Period: Period 1
Arm/Group | SPARC0921 | Placebo
Started (16 subjects were discontinued during Part 1 of the study.) | 392 | 0
Completed (6 subjects were discontinued during Part 3 of the study.) | 376 | 0
Not Completed | 16 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — MS related disease progression | 1 | 0
Not completed — Withdrawn | 1 | 0
Not completed — withdrew per sponsor | 1 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Did not meet eligibility criteria | 3 | 0
Period: Period 2
Arm/Group | SPARC0921 | Placebo
Started (80 subjects were discontinued in Part 2 of the study.) | 376 | 0
Completed | 296 | 0
Not Completed | 80 | 0
Not completed — Withdrawal by Subject | 23 | 0
Not completed — Adverse Event | 22 | 0
Not completed — no analysis | 10 | 0
Not completed — Lack of Efficacy | 8 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Sponsor's withdrawal | 7 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — dose change | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Did not meet eligibility criteria | 3 | 0
Period: Period 3
Arm/Group | SPARC0921 | Placebo
Started | 147 | 149
Randomization | 147 | 149
Completed | 146 | 144
Not Completed | 1 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — incorrect treatment | 0 | 1
Not completed — Sponsor's withdrawal | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects discontinued:
  During Part 1: 16 During Part 2: 80 During Part 3: 6 (5 in Placebo0921 and 1 subject in SPARC0921) Intent to treat population: 293 subjects (146 in Placebo0921 and 147 in SPARC0921)
Groups:
- SPARC0921: SPARC0921 Subjects who received SPARC0921 Dose Regimen I at Visit 1: 392 Received SPARC0921 Dose Regimen II at Visit 2 (Safety Population): 376 Randomized at Visit 7 to receive Dose Regimen III: 147
- Placebo0921: Placebo0921
  Randomized at Visit 7: 149
- Total: Total of all reporting groups
Arm/Group | SPARC0921 | Placebo0921 | Total
Number analyzed (Participants) | 147 | 146 | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (10.39) | 51.0 (9.39) | 49.9 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 99 | 204
  Male | 42 | 47 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 137 | 136 | 273
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 19 | 34
  White | 131 | 122 | 253
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure Rate
Description: Percentage of subjects who had treatment failure Clinical Global Impression of Change of ≥ 5 and at least one movement with ≥ 1 unit increase in modified Ashworth score from baseline.
  The modified Ashworth scale is a 6-point scale as follows: Minimum score of 0 (better outcome) = no increase in tone Maximum score of 4 (worst outcome) = affected part(s) rigid inflexion or extension.
  The clinician (other than the one performing the Modified Ashworth Scale assessment) rated his/her overall (global) impression of change in spasticity using the 7-point scale shown below: Minimum score of 1 (better outcome) = very much improved Maximum score of 7 (very much worse) = very much worse
Time Frame: Week 22
Population: Intent to treat population: SPARC0921, N=147 and and Placebo, N=146
Measure: Number; unit: percentage of subjects
Groups:
- SPARC0921: SPARC0921
- Placebo0921: Placebo0921
Arm/Group | SPARC0921 | Placebo0921
Number analyzed (Participants) | 147 | 146
percentage of subjects | 36.1 | 43.2
Statistical Analysis 1: Comparison: SPARC0921 vs Placebo0921; Test type: Superiority; p = 0.2062, Cochran-Mantel-Haenszel

2. Secondary Outcome: Severity of Spasticity Assessed by Subject Global Impression Severity Scale
Description: The subject was asked "Overall, how would you rate the severity of your spasticity over the past 24 hours?" The 7-point scale for Subject's global impression of severity assessment is as follows: minimum score of 1 = normal, no spasticity maximum score of 7 (worst outcome)= worst spasticity imaginable
Time Frame: Week 22
Population: Intent to treat population: SPARC0921, N=147 and Placebo0921, N=146
Measure: Number; unit: percentage of subjects
Groups:
- SPARC0921: Subject Global Impression of Severity of Spasticity in SPARC0921 group
- Placebo0921: Subject Global Impression of Severity of Spasticity in Placebo0921 group
Arm/Group | SPARC0921 | Placebo0921
Number analyzed (Participants) | 147 | 146
percentage of subjects
  Normal, no spasticity | 19.7 | 10.3
  Borderline spasticity | 6.8 | 13
  Mild spasticity | 26.5 | 20.5
  Moderate spasticity | 27.9 | 33.6
  Marked spasticity | 15.0 | 14.4
  Severe spasticity | 4.1 | 6.2
  Worst spasticity imaginable | 0 | 2.1
Statistical Analysis 1: Comparison: SPARC0921 vs Placebo0921; Test type: Superiority; p = 0.0485, Mantel Haenszel

ADVERSE EVENTS:
Time Frame: Week 22
Description: Part 2 and Part 3 safety data is displayed in the registry. Part A was a run-in period of the study.
Groups:
- SPARC0921- Part 3: SPARC0921 in randomized phase
- Placebo0921 - Part 3: Placebo0921 in randomized phase
- SPARC 0921 - Part 2: Open label
- Run-in Part 1: Open label run-in period
Arm/Group | SPARC0921- Part 3 | Placebo0921 - Part 3 | SPARC 0921 - Part 2 | Run-in Part 1
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/149 | 1/376 | 0/392
Serious Adverse Events (participants affected / at risk) | 3/147 | 0/149 | 12/376 | 0/392
Other Adverse Events (participants affected / at risk) | 23/147 | 25/149 | 226/376 | 6/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPARC0921- Part 3 (N=147) | Placebo0921 - Part 3 (N=149) | SPARC 0921 - Part 2 (N=376) | Run-in Part 1 (N=392)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 | 0
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
death (General disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPARC0921- Part 3 (N=147) | Placebo0921 - Part 3 (N=149) | SPARC 0921 - Part 2 (N=376) | Run-in Part 1 (N=392)
Muscle spasticity (Nervous system disorders) | 14 | 15 | 27 | 0
Headache (Nervous system disorders) | 6 | 4 | 14 | 0
Urinary tract infection (Infections and infestations) | 3 | 6 | 12 | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2 | 4 | 12 | 0
Blood pressure increased (Investigations) | 1 | 4 | 5 | 1
Fatigue (General disorders) | 4 | 0 | 24 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4 | 13 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 9 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 22 | 1
somnolence (Nervous system disorders) | 0 | 0 | 21 | 0
multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 12 | 0
dizziness (Nervous system disorders) | 0 | 0 | 10 | 1
Tremor (Nervous system disorders) | 0 | 0 | 6 | 0
vomitting (Gastrointestinal disorders) | 0 | 0 | 9 | 0
sinusitis (Infections and infestations) | 0 | 0 | 12 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 11 | 0
Oedema peripheral (General disorders) | 0 | 0 | 10 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 9 | 1
Asthenia (General disorders) | 0 | 0 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2012-02-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT01457352/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT01457352/SAP_001.pdf